CLINICAL TRIAL: NCT07119125
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Single and Multiple Dose Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MRT-8102 in Healthy Participants and in Participants at Cardiovascular Risk With Elevated CRP
Brief Title: A First-in-human, 3-part Study of MRT-8102 in Healthy Participants and Participants at Cardiovascular Risk With Elevated CRP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Monte Rosa Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRT-8102-001
Record Dates: First submitted 2025-07-30; First posted 2025-08-12 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers; Elevated CRP
Keywords: MRT-8102; MRT-8102-001; MRT; Monte Rosa Therapeutics; Healthy Volunteers; Single Ascending Dose; Multiple Ascending Dose; SAD; MAD; CRP; Cardiovascular Risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Single Ascending Dose (MRT-8102) (Experimental): Single Dose of MRT-8102
  Interventions: Drug: MRT-8102
- Part 1: Single Ascending Dose (Placebo) (Placebo Comparator): Single Dose of Placebo
  Interventions: Drug: Placebo
- Part 2: Multiple Ascending Dose (MRT-8102) (Experimental): 7-day Daily Dose of MRT-8102
  Interventions: Drug: MRT-8102
- Part 2: Multiple Ascending Dose (Placebo) (Placebo Comparator): 7-day Daily Dose of Placebo
  Interventions: Drug: Placebo
- Part 3: elevated CRP (MRT-8102) (Experimental): 28-day Daily Dose of MRT-8102
  Interventions: Drug: MRT-8102
- Part 3: elevated CRP (Placebo) (Placebo Comparator): 28-day Daily Dose of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MRT-8102 — Oral capsules
  Arms: Part 1: Single Ascending Dose (MRT-8102); Part 2: Multiple Ascending Dose (MRT-8102); Part 3: elevated CRP (MRT-8102)
Drug: Placebo — Oral capsules
  Arms: Part 1: Single Ascending Dose (Placebo); Part 2: Multiple Ascending Dose (Placebo); Part 3: elevated CRP (Placebo)

SUMMARY:
The principal aim of this study is to obtain safety and tolerability data when MRT-8102 is administered orally as single and multiple doses to healthy participants and participants at cardiovascular risk with elevated CRP. This information, together with the pharmacokinetic (PK) data, will help establish the dose and dosing regimen suitable for future studies.

The study drug, MRT-8102, is experimental. This is the first study in which MRT-8102 will be given to humans.

Part 1: Healthy participants will receive a single oral dose of MRT-8102 or placebo on Day 1

Part 2: Healthy participants will receive multiple oral doses of MRT-8102 or placebo for 7 consecutive days

Part 3: Participants at cardiovascular risk with elevated CRP will receive multiple oral doses of MRT-8102 or placebo for 28 consecutive days

DETAILED DESCRIPTION:
The purpose of this study is to:

* Learn about the safety and tolerability of single and multiple ascending oral doses of MRT-8102 in healthy adult participants
* Learn about the safety and tolerability of 28-day daily dosing of MRT-8102 in participants at cardiovascular risk with elevated CRP

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria (all parts)

* Healthy, adult, male or females 18-65 years of age
* Non-smoker who has not used nicotine- and tobacco -containing products for at least 3 months prior to start of study
* Able to swallow oral medications
* Abstain from caffeine- and methylxanthine-containing beverages or food

Parts 3: Inclusion Criteria

* Elevated CRP value ≥3.0 mg/L at the time of screening
* Evidence of cardiovascular risk factors
* No signs or symptoms of acute disease
* No ECG finding of clinical significance

Exclusion Criteria (All Parts)

* History or presence of clinically significant medical or psychiatric condition or disease
* Underwent surgical intervention or an operation withing 6 weeks prior to start of study
* Has active TB, latent TB, a history of TB, or had close contact with a person with active TB within 8 weeks prior to the first dosing
* Pregnant, breastfeeding, or planning a pregnancy or fathering a child during the study or within 3 months after the last study drug administration.
* Positive urine drug or alcohol screen results
* Positive results for human immunodeficiency virus (HIV), hepatitis B or Hepatitis C virus or history of resolved hepatitis
* Participation in another clinical study within 30 days or within 5 half-live (if known) prior to start of study
* Currently receiving other immunomodulators
* History of immunodeficiency, chronic inflammatory and chronic inflammation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single doses of MRT-8102 in healthy adult participants | 15 days
  Incidence of treatment-emergent adverse events by type severity seriousness and relationship to treatment and changes from baseline in safety-related clinical lab parameter, vital signs 12-lead ECGs and PEs
To evaluate the safety and tolerability of multiple ascending doses of MRT-8102 in healthy adult participants. | 21 days
  Incidence of treatment-emergent adverse events by type severity seriousness and relationship to treatment and changes from baseline in safety-related clinical lab parameter, vital signs 12-lead ECGs and PEs
To evaluate the safety and tolerability of 28-day daily dosing of MRT-8102 in participants at cardiovascular risk with elevated CRP | 56 days
  Incidence of treatment-emergent adverse events by type severity seriousness and relationship to treatment and changes from baseline in safety-related clinical lab parameter, vital signs 12-lead ECGs and PEs

SECONDARY OUTCOMES:
Characterize the PK Profile (peak plasma concentration) of MRT-8102 after single doses of MRT-8102 in healthy adult participants | Up to 8 days
  Peak plasma Concentration (Cmax)
Characterize the PK Profile (plasma concentration versus time) of MRT-8102 after single doses of MRT-8102 in healthy adult participants | Up to 8 days
  Area under the plasma concentration versus time (AUC)
Assess the effect of a high-fat/high-calorie meal on the PK (peak plasma concentration) of MRT-8102 02 in healthy adult participants | Up to 8 days
  Peak plasma Concentration (Cmax) - comparing fasted vs fed
Assess the effect of a high-fat/high-calorie meal on the PK (plasma concentration versus time) of MRT-8102 02 in healthy adult participants | Up to 8 days
  Area under the plasma concentration versus time (AUC) - comparing fasted vs fed
Characterize the PK profile (peak plasma concentration) of MRT-8102 in plasma after multiple doses of MRT-8102 in healthy adult participants | Up to 14 days
  Peak plasma Concentration (Cmax)
Characterize the PK profile (plasma concentration versus time) of MRT-8102 in plasma after multiple doses of MRT-8102 in healthy adult participants | Up to 14 days
  Area under the plasma concentration versus time (AUC)
Characterize the PK Profile (peak plasma concentration) of MRT-8102 when administered daily to participants at cardiovascular risk with elevated CRP | Up to 35 days
  Peak plasma Concentration (Cmax)
Characterize the PK Profile (plasma concentration versus time) of MRT-8102 when administered daily to participants at cardiovascular risk with elevated CRP | Up to 35 days
  Area under the plasma concentration versus time (AUC)
Assess the impact of MRT-8102 on serum concentration of CRP | Up to 35 days
  Mean changes from pre-dose baseline in serum CRP levels.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - ICON Clinical Research, Lenexa, Kansas
  - QPS, Springfield, Missouri
  - Endeavor Clinical Trials, San Antonio, Texas